CLINICAL TRIAL: NCT03090828
Title: Economic Evaluation of an Interactive Community-based Patient Education Platform Kidney Dialysis and Transplantation
Brief Title: Economic Evaluation of an Education Platform for Patients With End-stage Renal Disease
Acronym: PIC-R
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Centre Leon Berard (Other); Université Montpellier (Other); Telecom Bretagne (Unknown); Paris School of Economics (Unknown); Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: *P150958
Record Dates: First submitted 2017-02-20; First posted 2017-03-27 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-02

CONDITIONS: End-stage Renal Disease; Dialysis; Kidney Transplantation
Keywords: economic evaluation; e health
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (No Intervention): treatment as usual will be provided to patients
- app-based therapeutic education (Active Comparator): patients will have access to the app providing information of the disease as well as educational guidelines
  Interventions: Behavioral: app-based therapeutic education
- enhanced app-based therapeutic education (Experimental): patients will also have access to a chat room and discussion forum
  Interventions: Behavioral: enhanced app-based therapeutic education

INTERVENTIONS:
Behavioral: app-based therapeutic education — Patients will connect to a platform providing information on end-stage renal disease and to contact health care providers.
  Arms: app-based therapeutic education
Behavioral: enhanced app-based therapeutic education — Patients in the enhanced app group will also have access to a social network. (forum, chat room)
  Arms: enhanced app-based therapeutic education

SUMMARY:
1600 patients with severe, end stage renal disease or post transplant will be randomised 1:1:1 to either standard therapeutic education; or education using a specific app; or the enhanced interactive app using feedback messages.

The total follow up duration is 18 months. Primary endpoint is the cost utility of using app-based therapeutic intervention, secondary endpoints are: compliance with treatment guidelines, app use (professionals and patients), budget impact analysis

ELIGIBILITY:
Inclusion Criteria:

* severe end-stage renal disease Internet, literacy informed consent

Exclusion Criteria:

* did not fill the screening questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
cost utility, efficiency, budget impact | 18 months
  incremental cost utility ratio

SECONDARY OUTCOMES:
overall survival | 18 months
  percent of patients alive at 18 months
compliance and persistence | 18 months
  percent of patients using the app at 18 months
disease knowledge | 18 months
  answers to a questionnaire and change in the number of correct answers
lifestyle | 18 months
  changes in risk factors
app utilization by professionals and patients | 18 months
  number of connections, shares, likes
health care delivery organization | 18 months
  number of interactions (chats) between healthcare professionals and patients

IPD SHARING:
Plan to Share IPD: Undecided
JPAL plans to share the de-identified patient database

REFERENCES:
- [Derived] Pillebout E, Durand-Zaleski I, Farge L, Perrier L, de Chaisemartin C, Dupont JCK, Behaghel L, Rochaix L; Paris School of Economics and AP-HP Hospinnomics, Paris, France. Multicentre, randomised, economic evaluation of a web-based interactive education platform, simple or enhanced, for patients with end-stage renal disease: the PIC-R trial protocol. BMJ Open. 2022 Dec 9;12(12):e062613. doi: 10.1136/bmjopen-2022-062613. PMID 36600325